CLINICAL TRIAL: NCT07363902
Title: Clinical Safety and Feasibility Study for Non-CE Marked Medical Device: Evaluation of heepSync, a Novel Algorithm for Transcutaneous Electrical Stimulation of Respiratory Muscles in Mechanically Ventilated Patients.
Brief Title: Evaluation of heepSync, a Novel Algorithm for Transcutaneous Electrical Stimulation of Respiratory Muscles in Mechanically Ventilated Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tesai Care SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Heecap I
Record Dates: First submitted 2025-12-17; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ventilator-induced Diaphragm Dysfunction; VIDD; Weaning Failure
Keywords: Transcutaneous Electrical Stimulation; Mechanical ventilation; respiratory muscles

STUDY DESIGN:
Intervention Model Description: Multicenter Single Arm Pilot Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mechanical ventilated patients in ICU (Experimental): Single arm for device-treated patients
  Interventions: Device: Heecap

INTERVENTIONS:
Device: Heecap — Transcutaneous Electrical Stimulation of Respiratory Muscles

SUMMARY:
Up to 76% of ICU patients on mechanical ventilation develop significant respiratory muscle atrophy within the first 24 hours, contributing to prolonged ventilation, increased morbidity, and higher healthcare costs. To date, there is no practical, non-invasive technology that offers synchronized, personalized electrostimulation for both inspiratory and expiratory muscles during mechanical ventilation.

Heecap is a medical product designed to provide transcutaneous electrical stimulation of the respiratory muscles (TERM) that are involved in inspiration and expiration, detecting those in which it is clinically relevant and safe to provide such stimulation in assisted respiration.

The following study aims to evaluate the safety and preliminary performance of the stimulation algorithm in mechanically ventilated patients in the ICU. This evaluation will specifically focus on the algorithm's ability to synchronize stimulation with the patient's breathing patterns, and on evaluating the safety and feasibility of the TERM in activating respiratory muscles.

ELIGIBILITY:
Inclusion Criteria:

Patient population 1

* Adult patients with acute hypoxemic respiratory failure who have been under controlled mechanical ventilation for at least 24 hours prior to enrollment.
* Clinically stable: oxygen saturation > 90% with a fractional inspired oxygen ≤ 0.50, eternal PEEP ≤ 10 cm H2O, temperature ranging from 35.5 to 38.5 ºC, no intravenous administration of vasoactive agents.

Patient population 2

* Adult patients with acute hypoxemic respiratory failure who have been under pressure support mechanical ventilation for at least 24 hours prior to enrollment.
* Clinically stable: oxygen saturation > 90% with a fractional inspired oxygen ≤ 0.50, eternal PEEP ≤ 10 cm H2O, temperature ranging from 35.5 to 38.5 ºC, no intravenous administration of vasoactive agents.

Exclusion Criteria:

* Patients treated with neuromuscular blocking agents
* Patients with neuromuscular disease
* Patients with a pacemaker or past history of arrhythmia
* Patients with physical obstacles that prevent thoracic or abdominal electrostimulation (e.g., abdominal trauma, recent abdominal surgery, polytrauma, broken or irritated skin)
* BMI > 40 kg/m2
* Hemodynamically unstable (noradrenaline >0.1 microgram/kg/min)
* Pregnancy
* Patients under the age of 18
* The formalized ethical decision to withhold or withdraw life support
* Patient under guardianship
* Patients deprived of liberties
* Patients already enrolled in the present study, in a previous episode of acute respiratory failure.
* The patient who does not consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Device synchronization success rate | through study treatment phase completion (up to 3 days)
  Device feasibility in correctly stimulating breaths measured by the % of correct stimulated breaths of total breaths stimulated. All stimulated breaths will be analyzed and categorized as correctly stimulated or incorrectly stimulated.

SECONDARY OUTCOMES:
Incidence of AEs/SAEs | through study completion (up to 4 days)
  Number of Serious adverse events and Adverse events. Those will be collected and analyzed.
Transdiaphragmatic pressure (PDi) | During TERM on day 1 and day 2
  Comparison of PDi during stimulation session at day 1, stimulation session at day 2 and compared to basal (non stimulated, previous to session on day 1)
Muscle thickening fraccion | Day 1 and day 2 of treatment
  Difference of muscle thickening fraction in inspiration muscles and expiration muscles during stimulation (TERM sessions on day 1 and day 2) and compared to basal (pre-stimulation day 1)
Occlusion pressure (Pocc) | Day 1 and day 2
  Differences of Pocc mesured after stimulation sessions on day 1 and 2 and compared to basal (previous to stimulation session on day 1)

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitari de Vall d'Hebrón, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided